CLINICAL TRIAL: NCT00647361
Title: Short Term Effects of Neurally Adjusted Ventilatory Assist and Pressure Support Ventilation on Cardiac Performance
Brief Title: Mechanical Ventilation Controlled by the Electrical Activity of the Patient's Diaphragm - Effects on Cardiac Performance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Lukas Brander, MD, University Hospital - Inselspital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEK BE 217-06
Record Dates: First submitted 2008-03-19; First posted 2008-03-31 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Respiratory Failure; Cardiac Failure
Keywords: respiratory insufficiency; respiration; ventilators; diaphragm; electromyography; mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Heart Failure; Respiratory Aspiration | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NAVA (Experimental)
  Interventions: Device: Neurally adjusted ventilatory assist (NAVA) provided by a commercially available mechanical ventilator (Servo i, Maquet Critical Care, Solna, Sweden).

INTERVENTIONS:
Device: Neurally adjusted ventilatory assist (NAVA) provided by a commercially available mechanical ventilator (Servo i, Maquet Critical Care, Solna, Sweden). — Neurally adjusted ventilatory assist (NAVA) and pressure support ventilation (PSV)

SUMMARY:
Neurally adjusted ventilatory assist (NAVA) is a new concept of mechanical ventilation. NAVA delivers assist to spontaneous breathing based on the detection of the electrical activity of the diaphragm. We study the effect of NAVA on cardiac performance in critically ill, mechanically ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 - 85 years (extremes included)
2. Mechanical ventilation (tracheally intubated or tracheotomized)
3. Relevant interaction between the ventilator and the cardiac performance defined as an inspiratory deflection in central venous pressure or pulmonary diastolic pressure of ≥ 5 mmHg

   1. in 10 patients with impaired cardiac performance defined as either

      * a left ventricular ejection fraction of < 40% and/or
      * treatment with dobutamine ≥2μg/kg/min, or adrenaline ≥ 3μg/kg/min and/or
      * a cardiac index of ≤ 2.2 L•min-1•m2 and/or
      * a pulmonary artery occlusion pressure (PAOP) ≥ 18 mmHg
   2. in 10 patients with a history of chronic obstructive pulmonary disease (COPD) and delayed triggering-ON / cycling-OFF and/or evidence for wasted inspiratory efforts as evidenced by:

      * limitation of expiratory air flow and intrinsic PEEP as assessed by observation of the expiratory air flow curve and measurement of the airway pressure during an expiratory hold maneuver and/or
      * excessive activation of inspiratory and / or expiratory muscles as assessed by observation of the patient
4. Presence of a pulmonary artery catheter and an arterial pressure line
5. Subject itself or its next of kin has given written informed consent

Exclusion Criteria:

1. Patient is less than 18 years or more than 80 years of age
2. The attending physician refuses to allow enrollment
3. The patient refuses informed consent
4. Next of kin is unavailable or refuses informed consent
5. Pregnant or breast-feeding female. A pregnancy test will be performed in all female patients less than 60 years of age. The patient will not be enrolled in the study if the test result is positive.
6. Any contraindication to insertion/exchange a nasogastric tube, including (but not limited to): severe oropharyngeal malformation or bleeding; esophageal varices, tumor, infection, stenosis, or rupture
7. Presence or suspicion of diaphragm injury
8. Hemophilia or other severe bleeding disorder
9. Presence or suspicion of a central nervous system (CNS) disorder, including (but not limited to): CNS infarction, bleeding, tumor, or infection
10. History of heart and/or lung transplantation
11. Any mechanical cardiac assist device (including intraaortic balloon pump)
12. Any contraindication to reduce sedation or to stop neuromuscular blockage in order to allow spontaneous breathing
13. The patient needs to be ventilated with a mode of MV controlling for tidal volume or for airway pressure as per attending physician.
14. Severe hemodynamic instability as judged by the attending physician
15. Planned or anticipated intervention within the study period necessitating either transfer out of the ICU or requiring prolonged interaction with the patient.
16. a fraction of inspired oxygen (FiO2) of > 0.8
17. The patient currently participates in another interventional clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Cardiac stroke volume index. | end of experimental periods

SECONDARY OUTCOMES:
Global delivery of oxygen | end of experimental period

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Brander, MD, Principal Investigator — Department of Intensive Care Medicine, University Hospital - Inselspital, Bern, Switzerland
Locations (1):
- Department of Intensive Care Medicine, University Hospital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Sinderby C, Navalesi P, Beck J, Skrobik Y, Comtois N, Friberg S, Gottfried SB, Lindstrom L. Neural control of mechanical ventilation in respiratory failure. Nat Med. 1999 Dec;5(12):1433-6. doi: 10.1038/71012. No abstract available. PMID 10581089
- [Derived] Berger D, Bloechlinger S, Takala J, Sinderby C, Brander L. Heart-lung interactions during neurally adjusted ventilatory assist. Crit Care. 2014 Sep 12;18(5):499. doi: 10.1186/s13054-014-0499-8. PMID 25212533